CLINICAL TRIAL: NCT02413788
Title: Impact of Aerobic Training and Combined in Inflammatory Markers in Patients With Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Profa. Dra. Vera Lúcia dos Santos Alves, PhD in health sciences, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fcmscsp
Record Dates: First submitted 2015-03-31; First posted 2015-04-10 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2019-11

CONDITIONS: Scoliosis; Adolescent Scoliosis
Keywords: adolescent idiopathic scoliosis; inflammatory markers; exercise
MeSH Terms: conditions — Scoliosis; Motor Activity | interventions — Exercise; Exercise Test

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combined group (treadmill and resisted) (Experimental): - 10 minutes of warming, aerobic training 40 minutes on a treadmill (60-80% of maximum heart rate) and resisted training in equipment and free weights for 10 minutes with a set of 10 repetitions in quadriceps, triceps and biceps of the arms and legs (36 sessions)
  Interventions: Other: combined exercise; Device: treadmill
- aerobic group (treadmill) (Active Comparator): 10 minutes of warming, aerobic training 40 minutes on a treadmill (60-80% of maximum heart rate) for 36 sessions
  Interventions: Other: aerobic exercise; Device: treadmill

INTERVENTIONS:
Other: aerobic exercise — aerobic training 40 minutes on a treadmill (60-80% of maximum heart rate)
  Arms: aerobic group (treadmill)
Other: combined exercise — aerobic training 40 minutes on a treadmill (60-80% of maximum heart rate); resisted training in equipment and free weights for 10 minutes with a set of 10 repetitions in quadriceps, triceps and biceps of the arms and legs
  Arms: combined group (treadmill and resisted)
Device: treadmill

SUMMARY:
Inflammatory markers have been analyzed in several diseases of unknown etiology, in the expectation of increasing therapeutic perspectives. This possibility arises from the different levels of tissue injury with low-grade chronic inflammation that have been observed in studies in which the markers were not evaluated traditionally, and today have influenced clinical management.

The investigators aimed, therefore, to evaluate the inflammatory markers in patients with AIS before and after aerobic and combined exercise training.

DETAILED DESCRIPTION:
Inflammatory markers have not been evaluated in adolescent idiopathic scoliosis (AIS), but this deformity potentially involves various musculoskeletal structures permanently, which justifies the analysis. A low-grade chronic inflammation may be related to the lower capacity in exercise performance observed in this population, which must be stimulated to perform standardized physical activity.

ELIGIBILITY:
Inclusion Criteria:

* thoracic curvature ≥ 45 degrees
* indication for surgical treatment of spinal deformity
* absence of pulmonary, cardiac, articular or neurological disorder, atopic dermatitis and previous or current allergy
* agree part in the research with a assent statement and the person responsible with the consent form and informed

Exclusion Criteria:

* acknowledged chronic liver or kidney inflammatory disease
* use of corticosteroids, acetylsalicylic acid or other nonhormonal anti-inflammatory clinical or laboratorial evidence of infection
* severe obesity

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
interleukin 1 | change from baseline in interleukin 1 at 3 months
  Inflammatory Markers
interleukin 6 | change from baseline in interleukin 6 at 3 months
  Inflammatory Markers
interleukin 8 | change from baseline in interleukin 8 at 3 months
  Inflammatory Markers

SECONDARY OUTCOMES:
distance in six-minute walk test | change from baseline in distance at 3 months
  analysis of distance
oxygen saturation in six-minute walk test | change from baseline in oxygen saturation at 3 months
  analysis of oxygen saturation at end of test
systolic blood pressure in six-minute walk test | change from baseline in systolic blood pressure at 3 months
  analysis of systolic blood pressure at end of test
diastolic blood pressure in six-minute walk test | change from baseline in diastolic blood pressure at 3 months
  analysis of diastolic blood pressure at end of test
heart rate in six-minute walk test | change from baseline in heart rate at 3 months
  analysis of heart rate at end of test
respiratory frequency in six-minute walk test | change from baseline in respiratory frequency at 3 months
  analysis of respiratory frequency at end of test
Borg scale in six-minute walk test | change from baseline in Borg scale at 3 months
  analysis of Borg scale at end of test
forced vital capacity (FVC) | change from baseline at 3 months
  analyzed in liters or % of predicted of lung capacity variation from baseline at 3 months
maximal inspiratory pressure (MIP) | change from baseline at 3 months
  analysis of maximal inspiratory pressure variation (cmH2O)
maximal expiratory pressure (MEP) | change from baseline at 3 months
  analysis of maximal expiratory pressure variation (cmH2O)
peak expiratory flow | change from baseline at 3 months
  peak expiratory flow variation analysis in liters / minute (l/min)
forced expiratory volume in the first second (FEV1) | change from baseline at 3 months
  analyzed in liters or % of predicted of lung volume variation from baseline at 3 months
forced expiratory volume in the first second (FEV1) / forced vital capacity (FVC) | change from baseline at 3 months
  Analysis (%) of the relationship between FEV1 and FVC with variation from baseline at 3 months
FORCED EXPIRATORY FRACTION (FEF25-75%) | change from baseline at 3 months
  analyzed in milliliters (ml) of lung volume variation from baseline at 3 months
FORCED EXPIRATORY FRACTION (FEF25-75%) / forced vital capacity (FVC) | change from baseline at 3 months
  Analysis (%) of the relationship between FEV1 and FVC with variation from baseline at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa of Sao Paulo Medical School, São Paulo, Brazil

REFERENCES:
- [Derived] Xavier VB, Avanzi O, de Carvalho BDMC, Alves VLDS. Combined aerobic and resistance training improves respiratory and exercise outcomes more than aerobic training in adolescents with idiopathic scoliosis: a randomised trial. J Physiother. 2020 Jan;66(1):33-38. doi: 10.1016/j.jphys.2019.11.012. Epub 2019 Dec 16. PMID 31859153